CLINICAL TRIAL: NCT03558308
Title: The Effects of Computer Based Cognitive Rehabilitation on Executive Functions in Patients With Acquired Brain Injury in the Chronic Phase: A Pilot Study
Brief Title: CBCR for Executive Functions in Patients With ABI in the Chronic Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katrine Sværke (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Katrine Sværke, Bsc. Psychology, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-18006890
Record Dates: First submitted 2018-06-03; First posted 2018-06-15 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Acquired Brain Injury; Cognitive Symptom; Executive Dysfunction
MeSH Terms: conditions — Brain Injuries; Neurobehavioral Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients know that one of the conditions is a control-condition not expected to have significant clinical effects (required by the danish scientific committee), but they don't know which treatment condition they are randomised to. The outcome assessor is blind to the group allocation of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brain+ with clinical support (Experimental): Intervention: Computer based cognitive rehabilitation. This group will train with the programme 'Brain+' and receive continuous support from a clinician during the intervention period.
  Interventions: Behavioral: Computer based cognitive rehabilitation
- Cogmed with continuous support (Experimental): Intervention: computer based cognitive rehabilitation. This group will train with the programme 'Cogmed' and receive continuous support from a clinician during the intervention period.
  Interventions: Behavioral: Computer based cognitive rehabilitation
- Brain+ without support (Experimental): Intervention: computer based cognitive rehabilitation. This group will train with the programme 'Brain+' but receive no support during the intervention period.
  Interventions: Behavioral: Computer based cognitive rehabilitation
- Sham-training group (Sham Comparator): Intervention: Sham computerized gaming. This group will train computerized solitaire and other computerized games which are thought to be generally cognitive stimulating but with a very limit load on executive functions. This group will receive continuous support during the intervention period.
  Interventions: Other: Sham computerized gaming

INTERVENTIONS:
Behavioral: Computer based cognitive rehabilitation — Computer based cognitive rehabilitation is a supplementary computerized tool for cognitive rehabilitation design to train various cognitive functions. Many programmes are available. The current study investigates the effects on two such programmes on rehabilitation of executive functions in the chronic phase after acquired brain injury.
  Arms: Brain+ with clinical support; Brain+ without support; Cogmed with continuous support
Other: Sham computerized gaming — Sham training with generally stimulating computer-games
  Arms: Sham-training group

SUMMARY:
This study examines the effects of computerbased cognitive rehabilitation on executive functions in the chronic phase after acquired brain injury

DETAILED DESCRIPTION:
This study examines the effects of computerbased cognitive rehabilitation on executive functions in the chronic phase after acquired brain injury using two clinically developed programmes and one sham-intervention. Furthermore, the study consists of Groups that receives the computerized training both with and witouth support from a professional.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are able to give an informed consent both verbally and in writing
* Persons in the chronic phase after stroke or traumatic brain injury (more than one year post onset)
* Persons who score less than the 30. Percentile in one or more of the primary outcome measures outlined above.

Exclusion Criteria:

* Persons with neurodegenerative diseases
* Persons with diseases which can influence executive functions such as ADHD
* Persons who are motorically or cognitively unable to use a tablet and complete the CBCR-training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
PASAT | 3 seconds
  Paced auditory serial addition test, test of verbal working memory
Trail making test A+B | 5 minutes
  Trail test A: Test of visual attention, trail test B: Test of visual working memory and cognitive shifts

SECONDARY OUTCOMES:
SDMT | 90 seconds
  Symbol digit modalities test: Test of processing speed
Word fluency test | 1 min
  Test of verbal fluency
Digit span (WAIS-IV) | 5 minutes
  Test of verbal memory (forward) and working memory (backward)
Spatial span (WMS-III) | 5 minutes
  Test of visuospatial memory (forward) and visuospatial working memory (backward)
Stroop colour and word test | 3 minutes
  Test of inhibition
BNI-FS | 10 minutes
  Barrow Neurological Institute Fatigue Scale: Test of fatigue after brain injury
Quality of Life after Brain Injury (QOLIBRI) | 10 minutes
  Questionnaire about quality of life
Wordlist, Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 10 minutes
  Verbal memory test

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Mogensen, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- Center for Hjerneskade, Amager, København, Denmark

IPD SHARING:
Plan to Share IPD: Undecided